CLINICAL TRIAL: NCT01854320
Title: Acceptance-based Behavioral Treatment for Obesity: Maintenance and Mechanisms
Acronym: MYH-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Evan Forman, Principal Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK095069 (NIH)
Record Dates: First submitted 2013-05-14; First posted 2013-05-15 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Acceptance-based Treatment; Standard Behavioral Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Acceptance-based treatment (Experimental): Behavioral therapy for weight loss focusing on acceptance-based cognitive strategies and techniques.
  Interventions: Behavioral: Acceptance-based treatment
- Standard behavioral treatment (Active Comparator): Standard behavioral therapy for weight loss, the "gold standard" treatment.
  Interventions: Behavioral: Standard behavioral treatment

INTERVENTIONS:
Behavioral: Acceptance-based treatment
  Arms: Acceptance-based treatment
Behavioral: Standard behavioral treatment
  Arms: Standard behavioral treatment

SUMMARY:
The primary goal of this project is to determine if an innovative behavioral weight loss program that incorporates new developments from the field of behavior therapy produces superior weight control than standard behavioral treatment. A sample of 200 adults from the community are participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 70
* Have a BMI between 27-50
* Have the ability to engage in physical activity (i.e., can walk at least 2 blocks without stopping for rest).
* Agree to provide permission for the research team to regularly contact your physician throughout the study to share information on changes in your weight.
* Successfully complete all steps in the enrollment process

Exclusion Criteria:

* You have a medical condition or psychiatric condition that may limit your ability to comply with the behavioral recommendations of the program or pose a risk to you during weight loss.
* You are pregnant or plan to become pregnant in the next three years.
* Report recently beginning a course of or changing the dosage of prescription medications that can cause significant weight loss or weight gain.
* You are participating in or plan to participate in another weight loss program in the next three years.
* The research team identifies any factors that would render you potentially unable or unlikely to follow the protocol, or unable to benefit from it.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline - 2-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chabria R, Hagerman CJ, Crane N, Ehmann M, Knudsen FM, Brown KL, Forman E, Butryn ML. Racial disparities in the efficacy of traditional versus acceptance-based behavioral weight loss. Health Psychol. 2025 Jul 24:10.1037/hea0001537. doi: 10.1037/hea0001537. Online ahead of print. PMID 40705619
- [Derived] Crochiere RJ, Kerrigan SG, Lampe EW, Manasse SM, Crosby RD, Butryn ML, Forman EM. Is physical activity a risk or protective factor for subsequent dietary lapses among behavioral weight loss participants? Health Psychol. 2020 Mar;39(3):240-244. doi: 10.1037/hea0000839. Epub 2020 Jan 9. PMID 31916827
- [Derived] Godfrey KM, Schumacher LM, Butryn ML, Forman EM. Physical Activity Intentions and Behavior Mediate Treatment Response in an Acceptance-Based Weight Loss Intervention. Ann Behav Med. 2019 Nov 9;53(12):1009-1019. doi: 10.1093/abm/kaz011. PMID 30951589
- [Derived] Butryn ML, Call CC, Schumacher LM, Kerrigan SG, Forman EM. Time to Peak Weight Loss During Extended Behavioral Treatment. Obesity (Silver Spring). 2018 Apr;26(4):658-664. doi: 10.1002/oby.22127. Epub 2018 Feb 14. PMID 29442440
- [Derived] Butryn ML, Arigo D, Raggio GA, Kaufman AI, Kerrigan SG, Forman EM. Measuring the Ability to Tolerate Activity-Related Discomfort: Initial Validation of the Physical Activity Acceptance Questionnaire (PAAQ). J Phys Act Health. 2015 May;12(5):717-6. doi: 10.1123/jpah.2013-0338. Epub 2014 Aug 7. PMID 25106049